CLINICAL TRIAL: NCT04611230
Title: EpidemiologiCal POpulatioN STudy of SARS-CoV-2 in Lake CounTy, Illinois: CONTACT
Brief Title: A Study to Assess Infection Rate of Severe Acute Respiratory Syndrome - CoronaVirus 2 (SARS-CoV-2) and It's Affect on Quality of Life in Adult Volunteers in Lake County, Illinois
Acronym: CONTACT
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: H20-308
Record Dates: First submitted 2020-10-29; First posted 2020-11-02 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Severe Acute Respiratory Syndrome - CoronaVirus 2 (SARS-CoV-2)
Keywords: Severe acute respiratory syndrome - coronavirus 2; SARS-CoV-2; Coronavirus disease 2019; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Adult Volunteers (Low Risk Group): Volunteers with jobs that do not require close contact with (i.e., within 6 feet of) the general public or co-workers.
- Adult Volunteers (Medium - Low Risk Group): Volunteers with jobs that require in-frequent contact with (i.e., within 6 feet of) the general public or co-workers.
- Adult Volunteers (Medium - High Risk Group): Volunteers with jobs that require frequent contact with (i.e., within 6 feet of) the general public or co-workers.
- Adult Volunteers (High Risk Group): Volunteers with jobs that require frequent and/or close contact with (i.e., within 6 feet of) individuals with high potential for exposure to known or suspected sources of COVID-19.

SUMMARY:
Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Lung failure is the main cause of death related to COVID-19 infection. The main objective of this study is to assess infection of SARS-CoV-2 and how quality of life is affected in adult volunteers in Lake County, Illinois.

Volunteers will be recruited through digital advertisements and participants will be required to fill an online questionnaire. Upon consent, participants will be required to provide nasal swab and blood sample. Approximately 1250 adult volunteers living or working in Lake County, IL will be enrolled.

Participants will be followed for approximately 9 months and will be required to provide nasal swab and blood samples every 3 months and complete questionnaires every 2 weeks.

There may be higher treatment burden for participants in this trial. Participants will be monitored by medical assessments, blood tests and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Currently living or employed in Lake County, Illinois.
* Have regular access to computer, smartphone or tablet and sufficient internet access to connect to study platform.
* Willing and able to provide informed consent for collection of online data and of respiratory and blood specimens.
* Willing and able to follow the procedures of the study.
* Able to complete survey in English or Spanish.

Exclusion Criteria:

* Unable to provide informed consent.
* Unable to perform the requested study tasks and unable or unwilling to assign a proxy informant to complete the tasks.
* Hospitalized at the time of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult volunteers living or employed in Lake County, Illinois.
Sampling Method: Non-Probability Sample
Enrollment: 1007 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Evidence of Prior SARS-CoV-2 Infection | Baseline (Week 0)
  SARS-CoV-2 infection prior to enrollment is assessed by Immunoglobulin G (IgG) serology testing and/or self-reported diagnosis.
Percentage of Participants With Current SARS-CoV-2 Infection | Baseline (Week 0)
  SARS-CoV-2 active infection is assessed by polymerase chain reaction (PCR) testing.
Percentage of Participants With Incidence of SARS-CoV-2 Infection | Up to Approximately 9 months
  Incidence of SARS-CoV-2 Infection is assessed by positive PCR test, positive IgG serology test or COVID-19 diagnosis.

SECONDARY OUTCOMES:
Percentage of Participants With COVID-19 Hospitalization | Up to approximately 9 months
  Percentage of participants with COVID-19 hospitalization prior to enrollment will be recorded.
Percentage of Participants With Influenza and COVID-like Illness | Up to approximately 9 months
  Influenza and COVID-like illness is an indicator of potentially undiagnosed COVID-19 illness.
Time to Infection | Up to approximately 9 months
  The analysis for overall time-to-infection will be conducted using the Kaplan-Meier method.
Time to Symptom Onset | Up to approximately 9 months
  The analysis for overall time to symptom onset will be conducted using the Kaplan-Meier method.
Time to Symptom Resolution | Up to approximately 9 months
  The analysis for overall time to symptom resolution will be conducted using the Kaplan-Meier method.
Change in Quality of Life (QOL) | Up to approximately 9.5 months
  Change in quality of life is assessed through 5-level EQ-5D questionnaire (ED-5Q-5L)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Great Lakes Clinical Trials /ID# 224874, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sanchez-Solino O, Kilpatrick RD, Johnson C, Fang Y, Ye Y, Alami NN, Zarish K, Krueger WS, Dreyer N, Gray GC. Longitudinal Molecular and Serological Evidence of SARS-CoV-2 Infections and Vaccination Status: Community-Based Surveillance Study (CONTACT). Infect Dis Ther. 2024 Apr;13(4):633-645. doi: 10.1007/s40121-024-00923-4. Epub 2024 Mar 10. PMID 38461480
- [Derived] Kilpatrick RD, Sanchez-Solino O, Alami NN, Johnson C, Fang Y, Wegrzyn LR, Krueger WS, Ye Y, Dreyer N, Gray GC. EpidemiologiCal POpulatioN STudy of SARS-CoV-2 in Lake CounTy, Illinois (CONTACT): Methodology and Baseline Characteristics of a Community-Based Surveillance Study. Infect Dis Ther. 2022 Apr;11(2):899-911. doi: 10.1007/s40121-022-00593-0. Epub 2022 Feb 2. PMID 35107821
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=H20-308&Latitude=&Longitude=&LocationName=#additional-resources-section